CLINICAL TRIAL: NCT04131634
Title: A Phase II Trial of Stereotactic Ablative Radiation (SAbR) for Urothelial Cancer Patients With Progression While on Anti-PD-1/PD-L1 Immunotherapy
Brief Title: Stereotactic Ablative Radiation for Oligo-Progression of Urothelial Cancer
Acronym: SAbR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial has terminated due to changes in standard of care since its activation, which has led to poor accrual.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Aurelie Garant, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1506
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Urothelial Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAbR 6 measurable lesions (Experimental): PD-L1 assessment on biopsy of metastatic site (biopsy will be performed if no prior metastasis sample available)
  Interventions: Radiation: Stereotactic Ablative Radiation

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiation — A stereotactic relocalization system that relies upon stereoscopic radiographs, implanted fiducials, or near real-time CT based verification will be used.Investigators will have the discretion to choose from biologically equivalent dose levels using 1, 3 or 5 fractions. All active lesions need to be addressed by local therapy

SUMMARY:
To evaluate the benefit of SAbR for oligo-progressive metastatic urothelial cancer.

DETAILED DESCRIPTION:
Oligo-progressive urothelial cancer with limited disease burden and progression on an anti-PD-1/L1 immune checkpoint inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18-years-old
* ECOG performance status 0-2
* Patients must have pathology-proven metastatic urothelial carcinoma, with tissue sampling of at least the primary tumor. Tissue sampling of each presumed metastatic site is not necessary, provided that the patient already has a confirmed diagnosis of urothelial cancer.
* Patients must be on immune checkpoint inhibitor therapy with radiographic scans to verify oligo-progression of at least one and ≤ 6 sites of disease per RECIST 1.1.

  * Any of the currently FDA-approved PD-1/PD-L1 inhibitors are allowed. These include pembrolizumab, nivolumab, atezolizumab, avelumab, and durvalumab.
  * At least 1 metastatic lesion must show stable disease, partial response or complete response per RECIST 1.1.
* Patients must be able to understand and willing to sign written informed consent.
* Patients must have acceptable tolerability of ongoing therapy as decided by the treating medical oncologist.
* Patients must have a desire to continue ongoing therapy.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy, or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
  * Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Inability to receive further immune checkpoint inhibitor therapy
* Anticipated survival of fewer than 12 weeks
* Daily steroid requirement of > 10 mg prednisone or prednisone-equivalent. Steroid replacement therapy for adrenal insufficiency is permitted.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) at 6 months | 6 months
  Progression free survival (PFS) at 6 months in the patients for whom SAbR is added to the ICI after progression on ICI. PFS will be defined as the combination of progressive disease from SAbR start date and death from any cause.

SECONDARY OUTCOMES:
The disease control rate | 6 months
  The disease control rate in patients for whom SAbR is added to ICI after progression on ICI. DCR will be assessed per RECIST 1.1 criteria and defined as the combination of: Complete Response (CR), Partial Response (PR), or Stable Disease (SD).
The time to next-line systemic therapy | 6 months
  The time to initiation of next-line systemic therapy following the addition of SAbR to ICI after progression on ICI.
Overall survival of patients | 6 months
  The overall survival of patients since progression on ICI or at the study registration. Overall survival (OS) will be defined using the interval between enrollment and death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Aurelie Garant, Principal Investigator — University of Texas Medical Center
Locations (1):
- Aurelie Garant, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided